CLINICAL TRIAL: NCT05822505
Title: Prospective, Multicentre Study to Assess Performance of the Mpact 3D Metal MonoCer Cup Implant in Primary Total Hip Replacement
Brief Title: Monocer AOANJRR Registry-nested Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.026.001
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Survival, Prosthesis
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study titled "Prospective, Multicentre Study to Assess Performance of the MonoCer Acetabular Cup in Primary Total Hip Replacement" is a multi-centre prospective registry-nested cohort study, using AOANJRR's web-based data collection system integrated with Registry data collection, designed to assess the ten-year clinical outcome of the MonoCer Acetabular Cup in Primary Total Hip Replacement. The primary outcome measure is mortality and secondary measures are PROMs and complications.

DETAILED DESCRIPTION:
This study titled "Prospective, Multicentre Study to Assess Performance of the MonoCer Acetabular Cup in Primary Total Hip Replacement" is a multi-centre prospective registry-nested cohort study, using AOANJRR's web-based data collection system integrated with Registry data collection, designed to assess the ten-year clinical outcome of the MonoCer Acetabular Cup in Primary Total Hip Replacement. The primary outcome measure is mortality and secondary measures are PROMs and complications.

The purpose and objectives of this study are to assess and document the clinical outcomes in a group of primary total hip arthroplasty patients having this surgery for the management of end-stage osteoarthritis. Survivorship and changes in pain and function as well as death will be assessed. The design of this study will also allow, if required the continued follow-up after the initial 2 years to determine mid and long-term survivorship and performance of this cohort.

All patients will receive primary hip arthroplasty standard of care (pre and post operatively) as defined by each participating surgeon. In addition to the Medacta MonoCer Acetabular Cup. There shall be no investigational, experimental or "off-label" use of the device. There will be no experimental or investigational devices used. There will be no experimental or investigational surgical techniques used. The devices and products will be used in accordance with their instructions for use and/or approved labelling.

A prospective study will be conducted using the AOANJRR web-based data collection system (RAPID). Eligible and consented participants are registered in the RAPID system. The PROMs will be completed by patients via the RAPID system.

• Surgeons will determine patient eligibility, providing informed consent prior to enrolment and registration in RAPID.

Participating sites will send procedure data to the AOANJRR as per standard practice, this data is then linked to the study participant. All data will be stored in a secure data repository.

* A minimum of 280 patients will be recruited over an 18-month period.
* All data will be integrated with routinely collected Registry data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary total conventional hip replacement and are suitable for cementless acetabular cup according to the indications for use (On-label use).
* Use of the Medacta Mpact 3D Metal MonoCer acetabular cup prosthesis.
* Adults aged between 18 and 75 years at the time of registration.
* Ability to give informed consent.
* Patients who are informed of the conditions of the study and are willing to participate for the length of the prescribed follow-up period.

Exclusion Criteria:

Exclusion Criteria

* Rheumatoid arthritis.
* Patients with a history of active infection.
* Any case not described in the inclusion criteria.
* Revision procedures.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At least 280 patients will be recruited who will have the Mpact 3D Metal MonoCer acetabular cup prosthesis from four surgeons in Australia.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Survival rate at 2 years compared to all other acetabular cups utilising AOANJRR data revision rates. | 2 years
  Evaluation of MonoCer acetabular cup revision rates in comparison to all other TGA approved acetabular cup revision rates Analysis of reasons for revisions.
Survival rate at 5 years compared to all other acetabular cups utilising AOANJRR data revision rates. | 5 years
  Evaluation of MonoCer acetabular cup revision rates in comparison to all other TGA approved acetabular cup revision rates Analysis of reasons for revisions.
Survival rate at 10 years compared to all other acetabular cups utilising AOANJRR data revision rates. | 10 years
  Evaluation of MonoCer acetabular cup revision rates in comparison to all other TGA approved acetabular cup revision rates.
  Analysis of reasons for revisions.

SECONDARY OUTCOMES:
Collecting, assessing and documenting patient reported hip function, pain, pre-operative expectations and post-operative satisfaction with EQ-5D-5L | pre-op, 6 months, 1 year, 2 years, 5 years, 10 years
  Assessments / Questionnaires (Patient Reported Outcome Measures) EQ-5D-5L (EuroQol) min=0 (worst score) max=100 (best score) The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Collecting, assessing and documenting patient reported hip function, pain, pre-operative expectations and post-operative satisfaction with OHS | pre-op,6 months, 1 year, 2 years, 5 years, 10 years
  Assessments / Questionnaires (Patient Reported Outcome Measures) OHS
  The OHS is a short 12-item survey that can be done with pen and paper, or online.
  Patients are asked to reflect on their pain and functional ability over the previous four weeks. There are two domains (pain and function) with six items or questions in each. Each item has five possible responses. In the original scoring responses were from 1 = least difficult to 5= most difficult. Item scores are summed to give a total score from anywhere between 12 and 60. The lower the score, the better the outcome.
Collecting, assessing and documenting patient reported hip function, pain, pre-operative expectations and post-operative satisfaction with HOOS | pre-op,6 months, 1 year, 2 years, 5 years, 10 years
  Assessments / Questionnaires (Patient Reported Outcome Measures):
  HOOS
  HOOS: The hip disability and osteoarthritis outcome score (HOOS) is a questionnaire intended to be used to assess patient's opinion about their hip and associated problems, and to evaluate their symptoms and functional limitations during a therapeutic process. The HOOS questionnaire is a patient-administered self-report questionnaire and takes 7 to 10 minutes to complete. It is designed to be self-explanatory and user-friendly[1]. The HOOS includes 40 items with five possible responses, graded from 0 to 4 (0 points = worst possible score; 100 points = best possible score).
Collecting, assessing and documenting patient reported hip function, pain, pre-operative expectations and post-operative satisfaction with MONA | 6 months, 1 year, 2 years, 5 years, 10 years
  Assessments / Questionnaires (Patient Reported Outcome Measures):
  MONA (Melbourne Orthopaedic Noise assesment)
  MONA questionnaire, which has a high sensitivity for the detection of noises, concerning noise frequency and the quality of noise. Patients were asked if any noise had been heard from their hip joint at any time after surgery.
Collecting, assessing and documenting patient reported hip function, pain, pre-operative expectations and post-operative satisfaction with VAS | pre-op,6 months, 1 year, 2 years, 5 years, 10 years
  Assessments / Questionnaires (Patient Reported Outcome Measures):
  VAS (Visual Analog Scale) from 0 (worst) to 100 (best) score.
  The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between paints with similar conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jit Balakumar, Principal Investigator — Melbourne Orthopaedic Group
Locations (1):
- Melbourne Orthopaedic Group, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No